CLINICAL TRIAL: NCT00740584
Title: Assessment of Local Retention and Duration of Activity of SPL7013 Following Vaginal Application of 3% SPL7013 Gel (VivaGel) in Healthy Volunteers
Brief Title: Retention and Duration of Activity of SPL7013 (VivaGel®) After Vaginal Dosing.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Starpharma Pty Ltd (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPL7013-003; NIH contract HHSN266200500042C; DAIDS ES number 10730
Record Dates: First submitted 2008-08-21; First posted 2008-08-25 (Estimated); Results first posted 2012-08-14 (Estimated); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: HIV Infections; HSV-2 Genital Herpes
Keywords: Prevention
MeSH Terms: conditions — HIV Infections | interventions — astodrimer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open Label, only arm (Experimental): 3%w/w SPL7013 vaginal gel (VivaGel)
  Interventions: Drug: 3% SPL7013 Gel (VivaGel)

INTERVENTIONS:
Drug: 3% SPL7013 Gel (VivaGel) — A single application of VivaGel applied to the vagina on five separate occasions, each occasion separated by a minimum of 5 days.

SUMMARY:
To assess the retention and anti-viral activity (human immunodeficiency virus (HIV) and herpes simplex virus 2 (genital herpes, HSV-2) of SPL7013 in cervicovaginal samples taken up to 24 hours after administration of 3% SPL7013 in the vagina. There is no hypothesis for this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 18-45 with regular menstrual cycles, free from sexually transmitted infections and using adequate contraception

Exclusion Criteria:

* Any condition, including genital conditions, sexually transmitted infection, menopause, and/or allergies that would make the study participant unsuitable for the study.
* Pregnancy or breast-feeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-08; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Australia

REFERENCES:
- [Background] Price CF, Tyssen D, Sonza S, Davie A, Evans S, Lewis GR, Xia S, Spelman T, Hodsman P, Moench TR, Humberstone A, Paull JR, Tachedjian G. SPL7013 Gel (VivaGel(R)) retains potent HIV-1 and HSV-2 inhibitory activity following vaginal administration in humans. PLoS One. 2011;6(9):e24095. doi: 10.1371/journal.pone.0024095. Epub 2011 Sep 15. PMID 21935377

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 women recruited. Details to be provided in publication, which is in process.
Pre-assignment Details: Open label study, no assignment.
Period: Overall Study
Arm/Group | Open Label, Only Arm
Started | 12
Completed | 11
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open Label, Only Arm
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Number; unit: participants]
  Australia | 12

OUTCOME MEASURES:

1. Primary Outcome: HIV Antiviral Activity of Each of the Cervico-vaginal Samples (Samples Taken From the Vagina Using the Softcup)
Description: The HIV antiviral activity is the ability of each sample taken from the vagina (cervico-vaginal (CV) sample) to inhibit HIV virus from infecting a specific cell culture.
  The inhibition of HIV in the presence of the CV sample is compared to the inhibition of HIV in the cell culture with no CV sample added. This allows an assessment of the affect that the CV sample has.
Time Frame: at 3 hours
Measure: Median (Inter-Quartile Range); unit: percent anti-viral activity
Arm/Group | Open Label Active
Number analyzed (Participants) | 11
percent anti-viral activity | 96 (2) [95 to 98]

2. Secondary Outcome: Number of Participants With Adverse Experiences
Description: Number of participants with any untoward medical occurrence in a subject administered the Investigational Product, irrespective of any perceived causality to that study product
Time Frame: Approximately 13 weeks
Population: All Enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Open Label, Only Arm
Number analyzed (Participants) | 12
Participants | 7

ADVERSE EVENTS:
Arm/Group | Open Label, Only Arm
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label, Only Arm (N=12)
Related Genitourinary AEs (Reproductive system and breast disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No disclosure without SPL consent.